CLINICAL TRIAL: NCT06104943
Title: Stockholm hyperTRIglyceridemia REGister (STRIREG) Study
Acronym: STRIREG
Status: Active, not recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: K 2021-10399
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-09

CONDITIONS: Familial Hypertriglyceridemia
MeSH Terms: conditions — Hyperlipoproteinemia Type IV | interventions — Heredity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Index patients: All individuals who had had at least one plasma Triglyceride measurement between 1st January 2000 and 31st December 2021 at Karolinska University Laboratory or Unilabs AB in Stockholm County in Sweden.
  Interventions: Other: Heredity for cardiovascular disease; Other: Heredity for pancreatitis; Other: Heredity for type 2 diabetes; Other: Heredity for hypertriglyceridemia
- First degree relatives to index patients: Parents and the siblings to the index patients by interlinkage of personal identification numbers via the Swedish Multi-Generation register.

INTERVENTIONS:
Other: Heredity for cardiovascular disease — First degree relatives with a diagnosis of Cardiovascular disease.
  Groups: Index patients
Other: Heredity for pancreatitis — First degree relatives with a diagnosis of pancreatitis.
  Groups: Index patients
Other: Heredity for type 2 diabetes — First degree relatives with a diagnosis of type 2 diabetes.
  Groups: Index patients
Other: Heredity for hypertriglyceridemia — First degree relatives with hypertriglyceridemia
  Groups: Index patients

SUMMARY:
The STRIREG study is a retrospective longitudinal general population-based register study including all individuals who had had at least one plasma Tg measurement between 1st January 2000 and 31st December 2021 at Karolinska University Laboratory or Unilabs AB in Region Stockholm (population 2.41 million 2021). The exclusion criteria were a lack of a unique Swedish personal identification number (PIN). The index population consisted of 1,460,184 individuals between the age 0 and 107 years. The index population was extended to form the complete cohort (n=3,607,819) by associating the parents and the siblings (n=2,147,635) to the indexes by interlinkage of personal identification numbers via the Multi-Generation register (see below).

The study baseline for the index population was defined as the date for participant's first Tg measurement.

DETAILED DESCRIPTION:
Hypertriglyceridemia (hTG) is associated with atherosclerotic cardiovascular disease, pancreatitis, and non-alcoholic fatty liver disease in large population-based studies. Less is known about the impact on hereditary hTG and cardiometabolic disease status for the development of hTG and its associated cardiometabolic outcomes. hTG remains a target for lipid lowering therapies and with new pharmacological interventions being developed, there is a need to identify patients that will benefit most from treatment with these new medicines.

The population-based observational Stockholm hyperTRIglyceridemia REGister (STRIREG) study include 1,460,184 index individuals that have measured plasma triglycerides in the clinical routine in Region Stockholm, Sweden, between 1st January 2000 and 31st December 2021. The laboratory measurements also included basic haematology, blood lipid panel, liver function tests and HbA1c. Using the Swedish Multi-Generation register, 2,147,635 parents and siblings to the indexes were identified to form the complete study cohort. Laboratory data from participants were combined with data from several national registers that provided information on cause of death, medical diagnoses, dispensed medicines, and socioeconomic factors including country of birth, education level and marital status.

The multigenerational longitudinal STRIREG cohort provides a unique opportunity to investigate different aspects of familial hTG as well as heredity for other metabolic diseases. Important outcome measures include mortality, cardiovascular mortality, major cardiovascular events, development of incident diabetes, and non-alcoholic fatty liver disease. The STRIREG study will provide a deeper understanding of the impact of heredity on hTG and associated cardiometabolic complications.

ELIGIBILITY:
Inclusion Criteria: All individuals who had had at least one plasma Triglyceride measurement between 1st January 2000 and 31st December 2021 at Karolinska University Laboratory or Unilabs AB in Stockholm County Sweden.

Exclusion Criteria: No Swedish social security number.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Populationbased cohort originating from Stockholm County. with all individuals who had had at least one plasma Triglyceride measurement between 1st January 2000 and 31st December 2021 at Karolinska University Laboratory or Unilabs AB in Stockholm County Sweden. The first degree relatives are parents and siblings to the index patients identified through the Swedish Multi-Generation Register.
Sampling Method: Non-Probability Sample
Enrollment: 3607819 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Jan 1 2000 to Dec 31 2021
  All cause mortality
Cardiovascular mortality | Jan 1 2000 to Dec 31 2021
  Cardiovascular mortality
Pancreatitis | Jan 1 2000 to Dec 31 2021
  Pancreatitis
Major cardiovascular event (MACE) | Jan 1 2000 to Dec 31 2021
  Major cardiovascular event (MACE)

SECONDARY OUTCOMES:
Myocardial infarction | Jan 1 2000 to Dec 31 2021
  Myocardial infarction
Stroke | Jan 1 2000 to Dec 31 2021
  Stroke
Peripheral artery disease | Jan 1 2000 to Dec 31 2021
  Peripheral artery disease
Type 2 diabetes | Jan 1 2000 to Dec 31 2021
  Type 2 diabetes
Cardiac revascularization | Jan 1 2000 to Dec 31 2021
  Cardiac revascularization
Non alcoholic fatty liver disease | Jan 1 2000 to Dec 31 2021
  Non alcoholic fatty liver disease

IPD SHARING:
Plan to Share IPD: Undecided